CLINICAL TRIAL: NCT07215234
Title: A Phase 1/2, Study to Evaluate the Safety, Tolerability, and Efficacy of One-time Intravitreal Dose of SAR446597 in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Safety and Efficacy Study of a One-time Intravitreal Injection of SAR446597 in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DFI18231; 2025-524508-31 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-10-01; First posted 2025-10-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part I - SAR446597 open-label (OL) (Experimental): Participants will receive SAR at a dose specified for each cohort. Multiple dose levels of SAR446597 will be evaluated in successive cohorts of participants.
  Interventions: Drug: SAR446597
- Part II - SAR446597 Dose A (Experimental): Participants will receive SAR at a dose specified for each arm.
  Interventions: Drug: SAR446597
- Part II - SAR446597 Dose B (Experimental): Participants will receive SAR at a dose specified for each arm.
  Interventions: Drug: SAR446597
- Part II - Sham control (Sham Comparator): Participants will receive Sham at a dose specified for each arm.
  Interventions: Drug: Sham Comparator

INTERVENTIONS:
Drug: SAR446597 — Intravitreal injection
  Arms: Part I - SAR446597 open-label (OL); Part II - SAR446597 Dose A; Part II - SAR446597 Dose B
Drug: Sham Comparator — Sham periocular injection
  Arms: Part II - Sham control

SUMMARY:
This is a sequential Phase 1/2, two-part, multicenter study on safety, tolerability, and efficacy of one-time intravitreal SAR446597 for the treatment of participants with Geographic Atrophy (GA) secondary to Age-related Macular Degeneration (AMD).

The core phase duration will be approximately 2 years for each participant. An Extended Follow-Up (EFU) phase of 3 years follows the core phase.

The treatment is a one-time intravitreal injection of SAR446597 (or sham as applicable in Part II).

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or above
* Participants with diagnosis of GA secondary to age-related macular degeneration (AMD)
* Study eye with best corrected visual acuity (BCVA) ETDRS Snellen equivalent for dose escalation (Part I) between 20/40 and 20/320 and for expansion (Part II) equal or better than 20/200
* Study eye with GA lesion measuring between 2.5 and 17.5 mm2 for dose escalation (Part I) and between 2.5 and 14.0 mm2 for expansion (Part II). For multifocal disease, study eye with at least one single lesion of more than 1.25mm2 for both Part I and Part II

Exclusion Criteria:

* GA in the study eye caused by a disease different than AMD
* Presence of neovascularization or a history of treatment with an anti vascular endothelial growth factor agent in the study eye
* Any condition or treatment (ocular or systemic) or medical or surgical history in the study eye that may prevent visual acuity improvement or interfere with ocular safety or efficacy assessments
* Current or history of systemic complement targeting treatment in the past 12 months
* Use of ocular corticosteroids for 4 months (for ocular or periocular injections), 6 months (for intraocular implants) or 3 years (for long lasting intraocular implants) prior to screening in the study eye
* History of macular laser photocoagulation treatment, photodynamic- or thermotherapy or photo biomodulation in the study eye
* History of active ocular infection in the study eye in 6 months prior to screening
* Presence of active ocular or periocular infections
* Active uncontrolled glaucoma in the study eye
* History of uveitis or scleritis in either eye
* Previous gene therapy in either eye
* Any significant poorly controlled illness that would preclude study compliance and follow up

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-10-13 (Estimated); Study Completion 2032-07-22 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of ocular and non-ocular treatment-emergent adverse events (TEAEs) | Day 1 to Week 104
Incidence and severity of ocular and non-ocular treatment-emergent serious adverse events (TESAEs) | Day 1 to Week 104

SECONDARY OUTCOMES:
Change in square root-transformed (mm) and untransformed area (mm2) of GA | Baseline, Week 52, Week 104
Change in best-corrected visual acuity (BCVA) from baseline to Week 52 and Week 104 following SAR446597 administration measured with the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart | Baseline, Week 52, Week 104
Percentage of participants without loss of BCVA of ≥15 ETDRS letters from baseline in the study eye | Baseline, Week 52, Week 104
Incidence and severity of ocular and non-ocular TEAEs and TESAEs including clinically significant changes in safety parameters | Week 260 or End of Study

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Associated Retina Consultants - Peoria- Site Number : 8400011, Peoria, Arizona
  - Retina Macula Institute of Arizona- Site Number : 8400028, Scottsdale, Arizona
  - Vitreo Retinal Associates - Gainesville- Site Number : 8400004, Gainesville, Florida
  - University Retina - Lemont- Site Number : 8400005, Lemont, Illinois
  - The Retina Group of Washington - Chevy Chase- Site Number : 8400009, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants - Hagerstown- Site Number : 8400003, Hagerstown, Maryland
  - Oregon Retina- Site Number : 8400017, Eugene, Oregon
  - Mid Atlantic Retina- Site Number : 8400031, Bethlehem, Pennsylvania
  - Austin Clinical Research - Austin - Anderson Mill Road- Site Number : 8400007, Austin, Texas
  - Retina Foundation of the Southwest- Site Number : 8400001, Dallas, Texas
  - Texas Retina Associates - Dallas- Site Number : 8400006, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: DFI18231 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26880&tenant=MT_SNY_9011